CLINICAL TRIAL: NCT04198389
Title: Retrospective Clinical and Functional Evaluation of Patients Undergoing Knee Replacement With Small Implants
Acronym: SMALLIMPL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: I.R.C.C.S Ospedale Galeazzi-Sant'Ambrogio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMALLIMPLANTS
Record Dates: First submitted 2017-11-27; First posted 2019-12-13 (Actual); Last update posted 2019-12-13 (Actual); Status verified 2019-12

CONDITIONS: KNEE REPLACEMENT
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- partial knee replacement (Experimental): medial UNI, lateral UNI, patellofemoral replacement, combined UNI+ patellofemoral replacement, combined medial and lateral UNI
  Interventions: Procedure: PARTIAL KNEE REPLACEMENT

INTERVENTIONS:
Procedure: PARTIAL KNEE REPLACEMENT — PARTIAL KNEE REPLACEMENT

SUMMARY:
Retrospective evaluation of:

Functional results Clinical results Survivorship of knee replacement performed with small implants, isolated or combined

DETAILED DESCRIPTION:
Retrospective evaluation of partial knee replacements (medial UNI, lateral UNI, patellofemoral replacement, combined UNI+ patellofemoral replacement, combined medial and lateral UNI) performed in the Joint Replacement Department of the IRCCS Istituto Ortopedico Galeazzi.

evaluation includes: clinical examination, functional results, survivorship at 1, 2, 5 , 10 and 15 years.

ELIGIBILITY:
inclusion criteria:

* patients receiving medial UNI or lateral UNI or patellofemoral replacement or combined UNI+ patellofemoral replacement or combined medial and lateral UNI
* age > 18 years

exclusion criteria

* patients receiving total knee replacement
* patients having revision or a knee replacement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2017-07-20 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
KNEE SOCIETY SCORE | 2 years
  total scale range: 0 (minimum)-100 (maximum); excellent results: 80-100
KNEE SOCIETY SCORE | 5 years
  total scale range: 0 (minimum)-100 (maximum); excellent results: 80-100
KNEE SOCIETY SCORE | 10 years
  total scale range: 0 (minimum)-100 (maximum); excellent results: 80-100

CONTACTS AND LOCATIONS:
Locations (1):
- Irccs Istituto Ortopedico Galeazzi, Milan, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Romagnoli S, Vitale JA, Marullo M. Outcomes of lateral unicompartmental knee arthroplasty in post-traumatic osteoarthritis, a retrospective comparative study. Int Orthop. 2020 Nov;44(11):2321-2328. doi: 10.1007/s00264-020-04665-z. Epub 2020 Jun 20. PMID 32561964